CLINICAL TRIAL: NCT00835120
Title: Pioglitazone for the Treatment of Bipolar Disorder and Comorbid Metabolic Syndrome or Insulin Resistance
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other); Takeda Pharmaceuticals North America, Inc. (Industry)
Responsible Party: Principal Investigator, Joseph Calabrese, MD, Director, Mood Disorders Program, University Hospitals Cleveland Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-08-24
Record Dates: First submitted 2009-02-02; First posted 2009-02-03 (Estimated); Results first posted 2014-10-17 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2016-11

CONDITIONS: Metabolic Syndrome; Bipolar Depression; Insulin Resistance
MeSH Terms: conditions — Metabolic Syndrome; Bipolar Disorder; Insulin Resistance | interventions — Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pioglitazone (Experimental): Pioglitazone has been approved by the U.S. Food and Drug Administration (FDA) to help people who are diagnosed with diabetes
  Interventions: Drug: Pioglitazone

INTERVENTIONS:
Drug: Pioglitazone — An open-label 12-week trial of pioglitazone monotherapy. The investigators will titrate pioglitazone to the maximum tolerable dose up to 45mg per day.
  Other Names: Actos

SUMMARY:
The study is an open-label 8-week adjunctive trial of pioglitazone for the acute relief of bipolar depression comorbid with metabolic syndrome/insulin resistance. Subjects who experience a partial or full response will have the option of continuing in an acute continuation phase lasting up to 12 weeks. The extension phase will allow assessment of the safety and tolerability of pioglitazone during the acute continuation period.

ELIGIBILITY:
Inclusion Criteria:

* Be male or female between the ages of 18 and 70
* Diagnostic and Statistical Manual of Mental Disorders (DSM)-IV diagnosis of bipolar disorder (type I, II, or NOS)
* Currently depressed as confirmed by the MINI-Plus at the screening visit
* Currently receiving treatment with an anti-manic drug
* Meets criteria for metabolic syndrome or insulin resistance

Exclusion Criteria:

* Pregnancy or breast feeding
* Unstable or inadequately treated medical illness as judged by the investigator
* Severe personality disorder
* Serious suicidal risk
* Known history of intolerance or hypersensitivity to pioglitazone
* Treatment with pioglitazone in the 3 months prior to randomization
* Dependence on alcohol or drugs (other than nicotine) in the 3 months prior to study entry
* Currently taking an antidiabetic/glucose-lowering agent.
* Diagnosed with dementia
* Acute Mania as defined by a Young Mania Rating Scale (YMRS) score > 15
* Diagnosed with heart failure
* Transaminase elevation >2.5 times the upper limit of normal
* Presence of renal impairment (eg. creatinine > 1.5)
* Fasting blood glucose >150 mg/dL
* Hb A1c > 7.5%

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2009-03; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David E Kemp, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Kemp DE, Schinagle M, Gao K, Conroy C, Ganocy SJ, Ismail-Beigi F, Calabrese JR. PPAR-gamma agonism as a modulator of mood: proof-of-concept for pioglitazone in bipolar depression. CNS Drugs. 2014 Jun;28(6):571-81. doi: 10.1007/s40263-014-0158-2. PMID 24715548

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pioglitazone
Started | 34
Completed | 26
Not Completed | 8
Not completed — Lack of Efficacy | 1
Not completed — Lost to Follow-up | 3
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Pioglitazone
Number analyzed (Participants) | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.8 (10.9)
Gender [Count of Participants; unit: Participants]
  Female | 19
  Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 24
  More than one race | 0
  Unknown or Not Reported | 0
Bipolar Subtype [Number; unit: participants]
  Bipolar 1 | 27
  Bipolar 2 | 5
  Bipolar not otherwise specified | 2
Age of depression onset [Mean (Standard Deviation); unit: years] | 17.8 (10.9)
Age of mania/hypomania onset [Mean (Standard Deviation); unit: years] | 23.5 (19.2)
Age first treated for depression [Mean (Standard Deviation); unit: years] | 34.7 (11.3)
Age first treated for mania/hypomania [Mean (Standard Deviation); unit: years] | 40.8 (12.0)
Duration of mood state [Mean (Standard Deviation); unit: days] | 315.5 (331.6)
Number of prior hospitalizations [Mean (Standard Deviation); unit: hospitalizations] | 2 (4.0)
Number of prior suicide attempts [Mean (Standard Deviation); unit: suicide attempts] | 1.2 (2.0)
Employed [Number; unit: participants]
  Yes | 12
  No | 22
Medication treatment failures during current episode [Number; unit: participants]
  >=2 mood stabilizers (MS) or a MS + antidepressant | 26
  >=4 mood stabilizers or antidepressant | 15
Comorbid diagnoses [Number; unit: participants]
  Generalized anxiety disorder | 25
  Panic disorder | 11
  Post-traumatic stress disorder | 12
  Obsessive-compulsive disorder | 5
  Alcohol use disorder, lifetime | 19
History of physical abuse [Number; unit: participants]
  Yes | 10
  No | 24
History of verbal abuse [Number; unit: participants]
  Yes | 14
  No | 20
History of sexual abuse [Number; unit: participants]
  Yes | 9
  No | 25
Metabolic syndrome [Number; unit: participants]
  Yes | 32
  No | 2
Insulin resistance [Number; unit: participants]
  Yes | 30
  No | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in the Inventory of Depressive Symptomatology-Clinician Rated (IDS-CR) Score
Description: Inventory of Depressive Symptoms-Clinician rated, 30 item (IDS-C30) score change from baseline to study endpoint. IDS-C30 total scores can range from 0 to 84, with higher scores indicating a worse outcome
Time Frame: Week 0 - Week 8
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pioglitazone
Number analyzed (Participants) | 34
units on a scale | -16.5 (2.6)

2. Secondary Outcome: Change in Quick Inventory of Depressive Symptoms-Self Report (QIDS-SR16) Total Score
Description: The QIDS-SR16 is a 16-item, self report assessment. Total scores can range from 0 to 27, with higher scores indicating a worse outcome
Time Frame: Week 0 - Week 8
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pioglitazone
Number analyzed (Participants) | 34
units on a scale | -7.1 (1.2)

3. Secondary Outcome: Response Rates on the IDS-CR, Montgomery Asberg Depression Rating Scale (MADRS) and Quick Inventory of Depressive Symptomatology-Self-Report (QIDS-SR)
Description: A participant is considered to have responded if their total score on either the MADRS or QIDS-SR16 decreases by at least 50% between their Week 0 visit and Week 8 visit.
Time Frame: Week 0 - Week 8
Measure: Number; unit: participants
Arm/Group | Pioglitazone
Number analyzed (Participants) | 34
participants | 13

4. Secondary Outcome: Remission Rates Based on IDS-CR, QIDS-SR, and MADRS Scores
Description: A participant is considered in remission if their total score on the MADRS is > 7, their total score on the QIDS-SR16 > 6 and/or their total score on the IDS-CR is > 12 at Week 8.
Time Frame: Week 0 - Week 8
Measure: Number; unit: participants
Arm/Group | Pioglitazone
Number analyzed (Participants) | 34
participants | 8

5. Secondary Outcome: Change in Clinical Global Impressions-Bipolar Version (CGI-BP)
Description: The CGI-BP asks the clinician one question: "Considering your total clinical experience with this particular population, how mentally ill is the patient at this time?" which is rated on the following seven-point scale: 1=normal, not at all ill; 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; 7=among the most extremely ill patients.
Time Frame: Week 0 - Week 8
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pioglitazone
Number analyzed (Participants) | 34
units on a scale | -1.9 (0.3)

ADVERSE EVENTS:
Arm/Group | Pioglitazone
Serious Adverse Events (participants affected / at risk) | 0/34
Other Adverse Events (participants affected / at risk) | 16/34
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pioglitazone (N=34)
Dizziness (General disorders) | 4
Irritability (Psychiatric disorders) | 4
Increased Appetite (General disorders) | 4
Peripheral Edema (General disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes